CLINICAL TRIAL: NCT00042614
Title: Acute Cardiac Allograft Cellular Rejection and Cardiac Allograft Vasculopathy: Identification of Diagnostic Biomarkers and Target Pathways for Preventive Therapy
Brief Title: Study of Heart Transplant Rejection
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 020266; 02-CC-0266
Record Dates: First submitted 2002-08-01; First posted 2002-08-02 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-11-19

CONDITIONS: Heart Transplantation
Keywords: Genes; Heart; Lymphocytes; Proteomics; Transplant; Natural History; Heart Transplant; Healthy Volunteer; HV; Normal Control

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Controls: Matched to patients for age, gender and race
- Patients: Who have had heart transplants, awaiting, or controls screened.

SUMMARY:
This study will investigate the causes of acute and chronic rejection of transplanted hearts. To find better ways to detect, treat and possibly prevent heart transplant rejection, more information about the cause is needed. Acute and chronic heart transplant rejection may be caused by certain substances the body produces in response to the new heart. This study will try to find a blood or urine test that detects genes and proteins that can serve as markers of rejection. Such a test may lead to earlier detection and improved treatment.

Patients 18 years and above who are on a wait list for heart transplant at a UNOS-approved heart transplant center, whose institutional review board has approved this protocol, may be eligible for this study. Healthy volunteers will also be included in the study to establish a database of normal values for comparison with patients undergoing heart transplant. In addition, patients who have had a heart transplant within the past 1 to 5 years will be enrolled in a pilot study. Normal volunteers will be screened for participation with an electrocardiogram (EKG) and echocardiogram, non-invasive tests to evaluate heart function.

Participants will undergo the following procedures:

* Review of medical records Patients who have had a heart transplant and those on a wait list to receive a heart will have their medical records reviewed to collect information on their condition.
* Blood samples 60 cc (about 3 tablespoons) of blood will be collected from all participants by needle stick in a vein. The sample will be analyzed for genes and proteins that might predict heart rejection. In addition, many genes in blood cells and cells lining blood vessels that are unrelated to heart transplant rejection and whose functions or significance are unknown will also be examined for ideas for future research. Patients enrolled while on a wait list will, after transplantation, have an additional 44 cc (about 2 tablespoons) of blood collected at each heart biopsy and rejection episode during the first year of transplant, and 60 cc collected with each yearly biopsy for the next 9 years.
* Urine samples Between 100 and 300 cc (3 to 10 ounces) of urine may be collected from all participants to confirm blood test results

DETAILED DESCRIPTION:
Cardiac transplantation has been successful in improving survival in end stage heart failure. But graft rejection has limited survival after transplantation. In the first year, acute cellular rejection and infection remain the most common causes of morbidity and mortality. Afterwards, cardiac allograft vasculopathy (CAV), as a result of chronic vascular rejection, is the major cause of morbidity and mortality. Within the first year post-transplantation, almost two-thirds of recipients will experience at least one rejection episode. At five years post-transplantation, nearly 50% of survivors will have CAV. Clinically, the symptoms of acute rejection are relatively nonspecific (fatigue, dyspnea, fever). Most CAV patients remain asymptomatic until they develop serious problems such as myocardial infarction, heart failure, ventricular dysrhythmias or sudden cardiac death. Presently, the gold standard for diagnosing acute cardiac allograft rejection is right ventricular endomyocardial biopsy. This is an invasive method of diagnosis subject to morbidity and random sampling and interpretation error. Likewise, the gold standard for diagnosing CAV is cardiac catheterization with intravascular ultrasound, an invasive procedure also subject to morbidity. Noninvasive methods such as electrocardiography, echocardiography, and nuclear studies all have been studied, but have been unsuccessful, thus far, for either condition. Peripheral blood evaluations of cytokines and cytoimmunologic markers have also been unsuccessful in either condition. This clinical trial studies the feasibility of using functional genomics and proteomics to identify genes and proteins respectively that can serve as reliable biomarkers of acute cardiac cellular rejection and CAV. We plan to recruit subjects who are on the transplant waiting list. We will analyze the blood of these patients pre-transplant and serially post-transplant over one year and then regularly on a yearly basis. By correlating putative biomarkers with clinical, histological, and imaging based evidence of allograft disease we hope to build a database comprised of functional genomics, cytokine, cytoimmunologic and proteomics data relevant to the immunologic relationship between the donor organ and recipient. With this database we hope to obtain a minimal subset of differentially expressed genes, cytokines, cytoimmunologic and protein change profiles that is most predictive of both acute allograft rejection and CAV. This will eventually serve as the basis for a diagnostic blood test. Thus, with the application of functional genomics, cytokine, and cytoimmunologic analysis and proteomics we hope to derive a noninvasive method to detect both acute cellular cardiac allograft rejection and CAV, thereby minimizing the need for invasive methods of diagnosis. Further better understanding the genetic programs triggered and protein changes induced during rejection may lead to the identification of target pathways for developing new therapeutic approaches aimed at prevention.

Recently, several published reports have established that detection of donor DNA in recipient s blood can serve as a diagnostic tool of graft injury. The level of donor DNA measured as percentage of circulating cell-free donor DNA (%ccfdDNA) accurately diagnoses acute rejection with a high sensitivity and specificity, at times several months before the diagnosis by examining endomyocardial biopsies. The ability of cell free DNA to diagnose graft injury early opens a new window to re-examine markers of rejection. These markers are traditionally evaluated using biopsy results, often positive late during rejection. %ccfdDNA offers an opportunity to better characterize our analyses.

ELIGIBILITY:
* INCLUSION CRITERIA - for Transplant Patients:

  1. Adult heart transplant center generally accepts patients within the physiologic age range of 12 to 65 years old, however, for our study heart transplant patients must be 18 years of age or above.
  2. Indication for cardiac transplantation as outlined by the 24th Bethesda Conference on Cardiac Transplantation. These are as follows:
* Peak VO(2) less than 10 ml/kg per minute or less than 50% of maximal predicted VO(2) with achievement of anaerobic metabolism.
* Severe cardiac ischemia consistently limiting routine activity not amenable to surgical or percutaneous revascularization.
* Recurrent symptomatic ventricular arrhythmias refractory to all accepted therapeutic modalities.

EXCLUSION CRITERIA - for Transplant Patients:

Adult heart transplant centers exclude infants, toddlers, and children with a physiologic age less than 12, and adults with advanced physiologic age (less than 65), however, for our study we will exclude heart transplant patients less than 18 years of age.

The final decision to exclude a candidate from cardiac transplantation will be made by the hospital's heart transplant committee. The committee uses, as a guideline, the criteria outlined in the 24th Bethesda conference.

INCLUSION CRITERIA - for Control Subjects:

Any healthy normal man or women who is the appropriate age and gender for matching to a transplant patient.

EXCLUSION CRITERIA - For Control Subjects:

1. EKG with evidence of clinically relevant heart disease.
2. Echocardiogram with evidence of clinically relevant heart disease.
3. Any disease process that is not well controlled by medications.
4. Total tobacco use for greater than one month over the last 5 years.
5. Symptoms of coronary or cardiac insufficiency.
6. More than one major risk factor for coronary artery disease excluding gender or age.
7. Confirmed intrauterine pregnancy in women.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have had heart transplants, Patients Awaiting Heart Transplant, and Controls screened to obtain. Controls matched to patients for age, gender and race.@@@
Sampling Method: Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2003-04-07 (Actual)

PRIMARY OUTCOMES:
Rejection warranting medical intervention | end of study
  Medical intervention
Pathologically determined tissue rejection grades irrespective of treatment. | end of study
  Tissue Rejection

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Solomon, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Inova Fairfax Hospital, Falls Church, Virginia

REFERENCES:
- [Background] Zavazava N, Bottcher H, Ruchholtz WM. Soluble MHC class I antigens (sHLA) and anti-HLA antibodies in heart and kidney allograft recipients. Tissue Antigens. 1993 Jul;42(1):20-6. doi: 10.1111/j.1399-0039.1993.tb02161.x. PMID 8248891
- [Background] Pelletier RP, Morgan CJ, Sedmak DD, Miyake K, Kincade PW, Ferguson RM, Orosz CG. Analysis of inflammatory endothelial changes, including VCAM-1 expression, in murine cardiac grafts. Transplantation. 1993 Feb;55(2):315-20. doi: 10.1097/00007890-199302000-00017. PMID 7679529
- [Background] Herskowitz A, Mayne AE, Willoughby SB, Kanter K, Ansari AA. Patterns of myocardial cell adhesion molecule expression in human endomyocardial biopsies after cardiac transplantation. Induced ICAM-1 and VCAM-1 related to implantation and rejection. Am J Pathol. 1994 Nov;145(5):1082-94. PMID 7977640
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2002-CC-0266.html